CLINICAL TRIAL: NCT05067010
Title: Finding Retinal Biomarkers in Alzheimer's Disease
Acronym: FIREBALZ
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: D20170821
Record Dates: First submitted 2021-06-07; First posted 2021-10-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Biomarkers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Detailed ophthalmologic examination — * Visual acuity
  * Eye pressure measurement
  * Eye crystalline examination
  * Fundus examination
  * Optical coherence tomography of the retina
  * Retinophotos

SUMMARY:
CSF Alzheimer's disease (AD) biomarkers are the only one that reflect both Aβ and tau pathologies. There is increasing evidence for the presence of AD abnormalities in the retina of AD patients. Recent studies showed that they can be detected in living patients. Thus, retinal AD-linked abnormalities might be used as alternative diagnostic biomarkers for AD.

FIREBALZ study aims at identifying and validating retinal biomarkers for the diagnosis of Alzheimer's disease.

The study will include 160 patients in whom LP is indicated for assessment of CSF AD biomarkers according to French health authority (HAS) recommendations. Those patients will undergo a detailed neuro-ophtalmologic evaluation including retinal layers thickness evaluation (optical coherence tomography).

Univariate and multivariate analyses will be performed to test diagnostic properties of retinal parameters as compared to current diagnostic criteria including CSF biomarkers and logistic regression models will be used.

DETAILED DESCRIPTION:
Cerebrospinal fluid (CSF) Alzheimer's disease (AD) biomarkers are the only one that reflect both Aβ and tau pathologies. There is increasing evidence for the presence of AD abnormalities in the retina of AD patients. Recent studies showed that they can be detected in living patients. Thus, retinal AD-linked abnormalities might be used as alternative diagnostic biomarkers for AD.

FIREBALZ study aims at identifying and validating retinal biomarkers for the diagnosis of Alzheimer's disease.

The study will include 160 patients in whom lumbar puncture is indicated for assessment of CSF AD biomarkers according to French health authority recommendations. All patients will be recruited in the Cognitive Neurology Center (CMRR Paris Nord Ile-De-France), Paris, France. Patients will undergo a detailed neuro-ophtalmologic evaluation including complete ophthalmologic work-up to rule out chronic retinal pathology and retinal layers thickness evaluation (optical coherence tomography).

Inclusion period will be 40.5 months, Study duration for participants will be 6 at 12 weeks.

Two groups of patients will be defined for comparison according to LP results : patients with AD according to McKhann 2011 criteria and patients without AD Univariate and multivariate analyses will be performed to test diagnostic properties of retinal parameters and logistic regression models will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patient managed at the cognitive neurology center for cognitive impairment with a defined LP indication for the assessment of CSF AD biomarkers according to French National Health Agency recommandations in a clinical practice setting
* Patients with National Health Insurance coverage
* Patients willing to participate to the research and sign informed consent

Exclusion Criteria:

* Patient refusing to participate to research or unable to sign informed consent
* Patients without indication or displaying contraindication of LP
* Chronic retinal pathology interfering with analysis :

  * chronic glaucoma
  * diabetic retinopathy
  * severe hypertensive retinopathy
* Contraindication to brain MRI
* Other pathology considered as severe and impairing life expectancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients in whom lumbar puncture (LP) is indicated for assessment of CSF AD biomarkers according to French health authority (HAS) recommendations. All patients will be recruited in the Cognitive Neurology Center (CMRR Paris Nord Ile-De-France), Paris, France. Patients will undergo a detailed neuro-ophtalmologic evaluation including complete ophthalmologic work-up to rule out chronic retinal pathology and retinal layers thickness evaluation (optical coherence tomography).
  Inclusion period will be 40.5 months, Study duration for participants will be 6 at 12 weeks.
  Two groups of patients will be defined for comparison according to LP results : patients with AD (MCI and Dementia) according to McKhann 2011 criteria and patients without AD Univariate and multivariate analyses will be performed to test diagnostic properties of retinal parameters and logistic regression models will be used.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Diagnostic properties of retinal layers thickness measurement using OCT | up to 6 at 12 weeks
  Diagnostic properties of retinal layers thickness measurement using OCT for the diagnosis of probable AD according to McKahnn 2011 criteria combining clinical criteria and CSF biomarkers results.

SECONDARY OUTCOMES:
the diagnostic properties of optical coherence tomography (OCT) and retinophotos for the diagnosis of Alzheimer's disease | up to 6 at 12 weeks
  the diagnostic properties of optical coherence tomography (OCT) and retinophotos for the diagnosis of Alzheimer's disease
Relationship between retinal layer thickness measurments and retinal abnormalities | up to 6 at 12 weeks
  Relationship between retinal layer thickness measurments and retinal abnormalities
Relationship between retinal layer thickness measurments and markers of clinical | up to 6 at 12 weeks
  Relationship between retinal layer thickness measurments and markers of clinical
Relationship between retinal layer thickness measurments and imaging severity | up to 6 at 12 weeks
  Relationship between retinal layer thickness measurments and imaging (hippocampal volume and cortical atrophy evaluated semi-quantitatively on brain MRI) severity
the diagnostic properties of optical coherence tomography (OCT) and retinophotos for the diagnosis of cognitive alteration of neurodegenerative origin (all causes) | up to 6 at 12 weeks
  the diagnostic properties of optical coherence tomography (OCT) and retinophotos for the diagnosis of cognitive alteration of neurodegenerative origin (all causes)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COGNAT, Dr, Principal Investigator — Cognitive Neurology Center, CMRR Paris Nord Ile-De France
Locations (1):
- Centre Mémoire de Ressources et de Recherche Paris Nord, Paris, France

IPD SHARING:
Plan to Share IPD: No